CLINICAL TRIAL: NCT07283432
Title: Effect of Education Given With Virtual Reality Glasses on Self-Care Ability of Patients After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Tuba Yılmazer, Principal investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: bariatricsurgery
Record Dates: First submitted 2025-06-27; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bariatric Surgery; Virtual Reality; Education; Nursing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality group (Experimental): Patients in the experimental group will complete a "Patient Introduction Form" and a "Self-Care Ability Scale" the day before surgery. The researchers will also administer a "Simulator Illness Questionnaire" to determine their physiological status before the procedure. Before discharge from bariatric surgery, a 15-20 minute discharge training session will be provided using virtual reality headsets. The Simulator Illness Questionnaire will be repeated at the end of the procedure. The patient will be able to terminate the study at any time. Additionally, patients in the experimental group will receive counseling for 3 months. All patients in the experimental group will be asked about their Body Mass Index via telephone at 1 and 3 months after bariatric surgery and will complete the "Self-Care Ability Scale."
  Interventions: Device: virtual reality glasses
- Control (No Intervention): All patients in the control group will be asked to fill out the "Informed Consent Form" the day before the surgery and the "Self-Care Ability Scale" will be filled out by the researchers for the patients who agreed to participate in the study.
  No intervention will be applied to the control group patients and the clinic's routine practices will continue.
  All patients in the control group will be asked about their Body Mass Index via telephone interview at 1 and 3 months after bariatric surgery and the "Self-Care Ability Scale" will be filled out.

INTERVENTIONS:
Device: virtual reality glasses — Patients in the experimental group will be given 15-20 minutes of discharge training using virtual reality glasses before being discharged after bariatric surgery.
  Arms: Virtual reality group

SUMMARY:
This research aims to determine the effect of training given via virtual reality glasses on the self-care ability of patients after bariatric surgery. This study is a single-center, parallel-group, open-label, randomized controlled clinical trial. This study will be conducted with 60 patients who underwent colorectal surgery between August 2025 and December 2025. Participants will be randomized into two groups as the intervention group (n=30) and the control group (n=30). All patients in the experimental and control groups will be asked to fill out the "Informed Consent Form" and the "Self-Care Ability Scale" by the researchers on the day before the surgery, and the patients who agree to participate in the study will be given the "Patient Introduction Form" and "Self-Care Ability Scale" by the researchers. The "Simulator Illness Questionnaire" used in the Virtual Reality disease field will be applied to the patients in the experimental group, and their physiological conditions will be determined before the application. The patients in the experimental group will be given 15-20 minutes of discharge training with virtual reality glasses before being discharged after bariatric surgery. Watching videos with virtual reality glasses will be applied by the researcher in the patient rooms and beds. The Simulator Illness Questionnaire will be repeated at the end of the application. There will be no compelling effect that will negatively affect the health of the patients during the application, and the application will be terminated when the patients feel uncomfortable. A safe environment will be created so that there are no objects around the patients that they can bump into or trip over. The virtual reality glasses will be applied after a 5-10 minute trial period with the observer at the beginning. The patient can end the study at any time. If the patients use glasses/lenses, compliance will be checked. In addition, the patients in the experimental group will be counseled for 3 months.

The control group patients will not be subjected to intervention and the clinic's routine practices will continue.

All patients in the experimental and control groups will be asked about their Body Mass Index via telephone interviews at 1 and 3 months after bariatric surgery and the "Self-Care Ability Scale" will be filled out.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older, 65 years of age or younger,
* Who have undergone laparoscopic sleeve gastrectomy or laparoscopic gastric bypass surgery,
* Who have not developed any complications during or after the surgical procedure,
* Who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Patients who have not undergone laparoscopic surgery,
* Patients with neurological or psychological problems,
* Patients who have been transferred to the intensive care unit after surgery, - Emergency and unplanned cases,
* Patients diagnosed with cancer,
* Patients with visual, auditory or systemic disorders,
* Patients with balance problems,
* Patients diagnosed with hypertension and hypotension,
* Patients diagnosed with anxiety disorder or epilepsy will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Self-Care Abilities Scale | preoperative day 1, postoperative 1. month and postoperative 3. month
  The scale consists of 43 items. In our country, the scale was revised to 35 items. In the validity and reliability study of the scale, the Cronbach Alpha reliability coefficient was determined as 0.92.
  For the items containing statements about self-care abilities in the scale, there are the options "Does not describe me at all", "Does not describe me very much", "I have no idea", "Describes me a little" and "Describes me a lot". Each statement in the scale receives scores that can vary between zero and four. Reverse scoring is applied to the responses given to the eight items (3, 6, 9, 13, 19, 22, 26 and 31) containing negative expressions.
  The lowest score that can be obtained from the scale is zero, and the highest score is 140.
Simulator Sickness Questionnaire | postoperative day 4
  The Simulation Sickness Questionnaire (SSQ) is widely used to measure Virtual Reality illness. The simulator sickness questionnaire consists of 16 questions. These questions are located under 4 components: nausea (N), oculomotor (O), disorientation (D) and weighted total (T). The majority of studies conducted using the SSQ have reported only the Total Score score.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)